CLINICAL TRIAL: NCT04136509
Title: Biomaterials in the Surgical Rehabilitation of Oral and Maxillofacial Hard and Soft Tissue Defects
Brief Title: Microarchitecture of the Augmented Bone Following Sinus Elevation
Acronym: MAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Marton Kivovics, Senior lecturer, Semmelweis University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 52158-2/2015/EKU [0425/15]
Record Dates: First submitted 2019-10-16; First posted 2019-10-23 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-06

CONDITIONS: Alveolar Bone Loss; Sinus Pneumatization; Edentulous; Alveolar Process, Atrophy
Keywords: cone beam computed tomography (CBCT); microcomputed tomography (micro-CT); histomorphometry; sinus floor elevation; allograft; xenograft
MeSH Terms: conditions — Alveolar Bone Loss; Mouth, Edentulous; Atrophy | interventions — Sinus Floor Augmentation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The specialis tasked with histomorphometric, micro-CT and CBCT analysis has no knowledge on the intervention method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- allograft (Experimental): The filler used in sinus floor elevation is albumin impregnated allograft.
  Interventions: Procedure: sinus floor elevation; Procedure: bone core biopsy; Device: dental implant placement; Diagnostic Test: Cone Beam Computed Tomography scans (CBCT)
- xenograft (Experimental): The filler used in sinus floor elevation is anorganic bovine bone mineral.
  Interventions: Procedure: sinus floor elevation; Procedure: bone core biopsy; Device: dental implant placement; Diagnostic Test: Cone Beam Computed Tomography scans (CBCT)

INTERVENTIONS:
Procedure: sinus floor elevation — sinus floor elevation with the lateral technique
  Other Names: maxillary sinus augmentation
Procedure: bone core biopsy — After 6 month healing time reentry took place and bone core biopsy samples were collected from the augmented bone of the maxillary sinuses with a trephine drill. Biopsy samples were collected from the sites where the dental implants were to be placed.
Device: dental implant placement — During reentry after bone biopsy dental implants were placed.
Diagnostic Test: Cone Beam Computed Tomography scans (CBCT) — Preoperative CBCT scans are carried out before dental implant placement, 6 months after sinus floor elevations. Postoperative CBCT scans are taken 3 years after sinus floor augmentations.

SUMMARY:
In this prospective randomized clinical study sinus floor elevation procedures are preformed using different biomaterials with the lateral window technique. After a 6-month healing, at the time of dental implant placement bone core biopsy samples are harvested. The samples undergo micro-Ct and histomorphometric analysis.

DETAILED DESCRIPTION:
Aim of the study The aim of this prospective randomized study is to evaluate the remodeling capacity of albumin impregnated freeze-dried bone allograft in sinus floor augmentation by histomorphometry and micro-CT analysis and to compare it to anorganic bovine xenograft material.

Surgical methods Patients performed oral rinse with 0.2% chlorhexidine solution for 1 min before surgery. Under local anesthesia a full thickness flap was raised from a midcrestal incision along with two relieving incisions. Lateral window osteotomies were carried out with diamond burs. The Schneiderian membrane was carefully elevated. Bone graft material was packed in the defect with light force. Patients were randomly assigned to 2 groups based on the type of bone filler: albumin impregnated allograft (BoneAlbumin, OrthoSera GmbH, Krems an der Donau, Austria) or anorganic bovine bone mineral (ABBM), (Bio-Oss Geistlich Wolhusen, Switzerland). A porcine collagen membrane (Bio Gide, Geistlich GmbH, Wolhusen, Switzerland) was placed over the lateral window and fixed by titanium pins (Titan Pin Set, Ustomed Instruments Ulrich Storz GmbH & Co. KG, Tuttlingen, Germany). The buccal flap was mobilized to allow tension-free primary closure. The margins were stabilized with single interrupted sutures. Antibiotics (1 g amoxicillin-clavulanate twice a day for 5 days, or in case of side effects or known allergy to penicillin, 300 mg clindamycin 4 times a day for 4 days), anti-inflammatory drugs (50 mg diclofenac 3 times a day for 3 days), and chlorhexidine mouthwash (twice a day for 21 days from the first day after surgery) were prescribed. Sutures were removed after 10 days. After 6 months healing surgical re-entry procedure took place under local anesthesia. A bone core biopsy was taken with a trephine with an external diameter of 3.5 mm and an internal diameter of 2.5 mm (330 205 486 001 025 Hager & Meisinger GmbH, Neuss, Germany) and implants of at least 4.0 mm of diameter were placed into the grafted alveolus nonsubmerged.

Histomorphometry Bone core biopsy material was fixed in 10% buffered formaldehyde solution. Following decalcination and dehydration, the biopsy material was embedded in paraffin and 20 µm sections were prepared. The sections were stained with routine haematoxylin eosin stain. Sections were evaluated under a light microscope in magnification 40×-400× .

Histomorphometric measurements were completed on sections with Panoramic Viewer 1.15 (3DHISTECH Ltd., Budapest, Hungary) using a combination of Adobe PhotoShop (Adobe System Inc., San Jose, CA, USA) and ImageJ, the public domain NIH Image program (US National Institutes of Health' http://rsb.info.nih.gov/nih-image/) at 150× magnification. Two slides of the augmented areas in each bone core biopsy sample were evaluated to record area percentage of newly formed bone, residual particles of the bone graft material, and the bone marrow space according to published protocols. Histomorphometric data consisted of the area percentage of newly formed bone, residual particles of the graft material and bone marrow were identified in each section.

Micro-CT analysis The bone core biopsy samples were scanned using a microcomputed tomography (μCT) scanner (Skyscan 1172 X-ray microtomograph, Bruker µCT, Kontich, Belgium). After the acquisition, raw images were reconstructed using NRecon software (v.1.7.1.6., Bruker µCT, Kontich, Belgium). The morphometric variables relevant to our study calculated by CTAn software (v.1.17.7.2, Bruker µCT, Kontich, Belgium). On the reconstructed images of each sample the demarcation plane of the host and the augmented area was identified and the complete available tissue (maxilla or augmented bone, respectively) were selected as regions of interest (ROIs) for quantitative analysis.

Micromorphometric data was collected by evaluation of the augmented bone of the test or control group. Additional micromorphometric data was recorded by analyzing the native bone of the alveolar ridge within the bone core biopsy samples of both test and control group. The microarchitectural parameters of the augmented bone of the BoneAlbumin group and the ABBM group; the augmented bone of the BoneAlbumin group and the native bone of the alveolar ridge; the augmented bone of the ABBM group and the native bone of the alveolar ridge were compared.

Statistical analysis Percentage values of each bone core biopsy sample were used to calculate descriptive statistics for the histomorphometrical and quantitative µCT analysis. The results were analyzed statistically using the IBM SPSS Statistics 23 data analysis software program (IBM Corporation, New York, NY. USA). The Kruskal Wallis One-way ANOVA test was used to compare two sets of data for the statistical analysis of the histomorphometric results. One-way ANOVA test was used to compare three sets of data for the statistical analysis of the micromorphometric results of the micro-CT. Values of p < 0.05 were considered statistically significant.

CBCT CBCT imaging (PaX-Reve3D, Vatech, Hwaseong, South-Korea) was carried out prior to sinus floor elevation to evaluate the anatomy and possible pathology of the maxillary sinuses, then 6 months after bone augmentation prior to implant placement (preoperative CBCT), and 3 years after implant placement (postoperative CBCT). To register the preoperative and postoperative CBCT data by anatomical landmarks 3DSlicer 4.10.2 software (The Brigham and Women's Hospital, Inc. Boston, USA) was used. The ROIs were identified by determining the central axis of the implants and placing a virtual cylinder on the preoperative CBCT image sequence with a diameter of 2,5 mm and the length of 8 mm on this axis corresponding with the inner dimensions of the trephine used for bone core biopsy harvesting. The image sequences of selected ROIs were imported in CTAn software (v.1.17.7.2, Bruker micro-CT, Kontich, Belgium) and micromorphometric variables were calculated by the software.

Statistical analysis of CBCT results Correlation of the micromorphometric data obtained from the CBCT images and micro-CT images was determined by The Spearman's rank-order correlation. Statistical analysis was performed using the IBM SPSS Statistics 25 data analysis software program (IBM Corporation, New York, USA). Values of P < 0.05 were considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Periodontally healthy patients
* Edentulous posterior maxilla

Exclusion Criteria:

* History of systemic diseases, that alter bone metabolism (osteoporosis, diabetes mellitus),
* History of medication known to alter bone remodelling (bisphosphonates, RANK ligand inhibitor monoclonal antibodies, corticosteroids),
* History of uncontrolled medical or psychiatric disorders,
* Inflammations of the paranasal sinuses or the alveolar process,
* History of tumours or irradiation therapy in the head and neck region,
* Unwillingness to return for follow-ups,
* Pregnancy,
* Smoking,
* Inability to preform proper oral hygiene.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
newly formed bone percentage | 6 months
  newly formed bone area compared to total area in histomorphometry
BV/TV bone volume fraction | 6 months
  bone volume compared to total volume in micro-CT reconstruction

SECONDARY OUTCOMES:
bone gain | 3 years
  volume of augmented bone on CBCTs

CONTACTS AND LOCATIONS:
Overall Officials: György Szabó, Md PhD Msc, Study Director — Department of Oro-Maxillofacial Surgery and Stomatology Semmelweis University
Locations (1):
- Semmelweis University Department of Community Dentistry, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No